CLINICAL TRIAL: NCT01863264
Title: A Pilot Study on The Effects of Cold Liquids on the Pharyngeal Swallow in Preterm Infants With Dysphagia.
Brief Title: The Effects of Cold Liquids on the Swallowing Mechanism in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 460111-3
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Dysphagia
Keywords: dysphagia; swallowing; infant; premature; neonate; thermal; cold; bolus; temperature; deglutition; NICU; bottle; nippling
MeSH Terms: conditions — Deglutition Disorders; Premature Birth; Common Cold | interventions — Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cold Thin Liquid Barium (Experimental): Poland Spring Natural Spring Water will be placed in a refrigerator set to 36 °F, this will allow the water to cool to approximately 4-9 °C. As described by several authors, these waters will be used to mix the barium powder (Varibar® Thin Liquid Barium Sulfate for Suspension) to create a thin liquid consistency, with 50% dilution, which is found to be most similar to human milk and infant formula.
  the infant will be required to swallow 5 boluses of this cold liquid barium while bottle feeding.
  Interventions: Other: Cold Thin Liquid Barium

INTERVENTIONS:
Other: Cold Thin Liquid Barium — Cold thin liquid barium will be fed to the participant from a standard bottle (60ml Similac® Volu-Feeder® with an attached Similac® Infant Nipple and Ring (standard flow)). For this study the refrigerated (cold) thin liquid barium will be measured for an exact temperature of 4-9°C prior to administration to control for any temperature variation. A total of 5 swallows will be visualized and saved electronically on the hospital's electronic storage system.
  Other Names: Varibar® Thin Liquid Barium Sulfate for Suspension

SUMMARY:
The purpose of this study is to see if cold liquids improve the swallowing mechanisms in premature infants with swallowing difficulties (dysphagia). The only way to objectively diagnose dysphagia is by having that infant undergo a Video Fluoroscopic Swallow Study (VFSS), which allows direct visualization of the liquid bolus (barium) in real time. Infants suspected of having dysphagia and who are referred for a VFSS will be recruited for this study. Once consented, the infant will undergo a standard VFSS. If that infant is diagnosed with dysphagia, the study protocol will begin by keeping the infant the same position and feeding them cold liquid barium from an identical bottle. A total of 5 swallows will be visualized, which adds approximately 5-10 seconds to the study. Both the standard swallows and the study swallows will be recorded for analysis and comparison. It is hypothesized that the study swallows will have less deficits than the standard swallows. If an infant's standard VFSS does not indicate dysphagia, that infant will no longer be eligible for this study.

DETAILED DESCRIPTION:
Swallowing is a complex task that takes place in the mouth and throat. It involves tiny receptors that gather sensory information about the liquid. Those receptors send a sensory message to the brain, where it is processed. The brain then sends back motor messages to the muscles in the throat regarding what kind of motor movements to do in order to swallow that liquid safely. The motor movements must be carefully timed and coordinated to safely swallow the liquid with out it going near, or into the lungs. When the liquid goes down the wrong tube, or into the lungs, it is called aspiration.

Some infants that are born prematurely end up with swallowing problems when drinking from a bottle. This problem can lead to liquid, such as formula or breastmilk, to be aspirated. This is due to the infant's poor coordination of all the muscles needed to safely swallow.

Researchers have found that changing the sensory characteristics of the liquid alters the motor movements of the swallow. This is because the sensory receptors respond differently to different types if liquids. Studies using adults with swallowing problems has shown that swallowing cold liquids improves some of the swallowing difficulties. Based off of these observations, there are currently several therapies used in Neonatal Intensive Care Units (NICU) nationwide which use cold stimulation to improve swallowing in prematurely born infants, although, there has been no research studies proving it actually works.

The purpose of this study is to assess the effect of cold liquid on the swallow mechanism in preterm infants with swallowing difficulties. A video x-ray procedure, called a Videofluoroscopic Swallow Study (VFSS), is considered the gold standard when assessing the motor movements present in the throat when swallowing. The standard procedure for an infant VFSS involves bottle feeding room temperature liquid barium while looking at the swallow movements obtained from the video x-ray images. After consent is obtained, infants who are assumed to have swallowing difficulties will undergo a "standard" VFSS. If during the study they are found to have swallowing problems, the study protocol will then begin by introducing cold liquid barium from an identical bottle. A total of 5 swallows will be looked at and recorded for review at a later time. The standard procedure for that infant's VFSS will then continue.

The hypothesis is that cold liquids will improve the swallowing movements in premature infants with swallowing difficulty. Information gathered will support the use of cold liquids and cold stimulation in NICUs to help benefit these infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants born prematurely, as defined by birth at less than 37 weeks gestational age, referred for a videofluoroscopic swallow study (VFSS) due to suspected pharyngeal phase dysphagia.

Exclusion Criteria:

* Infants born prematurely with a corrected gestational age of 43 weeks or greater.

Max Age: 43 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pharyngeal Swallow Trigger | <2seconds post swallow trigger
  the interval in seconds between the first frame showing barium passing the posterior tongue to the first frame showing laryngeal elevation.
Laryngeal Penetration, Mild | <2 seconds post swallow trigger
  the occurrence of barium underneath the epiglottis, remaining in the upper 1/3 quadrant of the laryngeal vestibule
Laryngeal Penetration, Deep | <2 seconds post swallow trigger
  the occurrence of barium underneath the epiglottis, in the laryngeal vestibule to the level of the vocal folds
Tracheal Aspiration | <5 seconds post swallow trigger
  the occurrence of barium below the level of the true vocal cords
Nasopharyngeal Reflux | <2 seconds post swallow trigger
  the occurrence of barium detected in the nasopharynx, posterior or superior to the velum

SECONDARY OUTCOMES:
Pharyngeal residue | <5 seconds post swallow trigger
  the presence of residual barium coating the pharyngeal walls, pooling in the vallecula or pyriform sinuses post swallow (absent/mild/severe).
Silent Aspiration | <5 seconds post swallow trigger
  occurrence of a cough in the presence of aspiration (present/absent)
Laryngeal Clearance | <5 seconds post swallow trigger
  ability to clear larynx during penetration events (sufficient/insufficient)
Tracheal Clearance | <5 seconds post swallow trigger
  ability to clear trachea during aspiration events (sufficient/insufficient)

CONTACTS AND LOCATIONS:
Overall Officials: Louisa Ferrara, MS, CCC-SLP, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States